CLINICAL TRIAL: NCT05864937
Title: Comparison of Two Preventive Treatments for Patients With Recurrent Miscarriages Carrying a C677T Methylenetetrahydrofolate Reductase Mutation: 5-year Experience
Brief Title: C677T Methylenetetrahydrofolate Reductase Mutation
Acronym: C677T
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0045
Record Dates: First submitted 2018-08-23; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2018-09

CONDITIONS: Mutation
Keywords: recurrent miscarriages; aspirin; folic acid
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: infertily evaluation — All couples had undergone a standard infertility evaluation, which included medical history, physical examination, and assessment of tubal patency by either hysterosalpingography or laparoscopy and hormonal analysis on cycle day 3. A transvaginal ultrasound scan was performed on the second day of the cycle. On the same day, ovarian stimulation was carried out with recombinant FSH follitropin);rFSH;Gonal-F,MerckSerono,France,orfollitropin ; Puregon, MSD, France), urinary FSH (urofollitropin, Fostimon, France),orhMG(menotropin,Menopur,France)atastarting dose of 75 IU/day from the second day of the cycle.

SUMMARY:
To investigate the effect of anticoagulant treatment on pregnancy outcomes in patients with previous recurrent miscarriages (RM) who carry a methylenetetrahydrofolate reductase (MTHFR) gene mutation.

In this longitudinal retrospective study, patients with RM were treated during pregnancy with either: (i) 100 mg/day aspirin and 5 mg/day folic acid (group 1); or the same protocol plus 0.4 mg/day enoxaparin (group 2). An age-matched group of triparous women without RM or thrombophilia was used as the control group (group 3).

DETAILED DESCRIPTION:
Recurrent miscarriage (RM) is defined as three or more consecutive spontaneous fetal losses and it affects 0.3% to 1% of pregnancies.To investigate the effect of anticoagulant treatment on pregnancy outcomes in patients with previous recurrent miscarriages (RM) who carry a methylenetetrahydrofolate reductase (MTHFR) gene mutation.

In this longitudinal retrospective study, patients with RM were treated during pregnancy with either: (i) 100 mg/day aspirin and 5 mg/day folic acid (group 1); or the same protocol plus 0.4 mg/day enoxaparin (group 2). An age-matched group of triparous women without RM or thrombophilia was used as the control group (group 3).

ELIGIBILITY:
Inclusion Criteria:

* patients with three or more consecutive first-trimester miscarriage
* Three or more consecutive first-trimester miscatrriages
* C677T MTHFR gene mutation

Exclusion Criteria:

* Patients with the A1298C polymorphism

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with three or more consecutive first-trimester miscarriages who were carrying the C677T MTHFR gene mutation and were treated and followed-up by the Department of Obstetrics, Gynaecology and Reproductive Medicine, Amiens University Medical Centre, Amiens, France between January 2006 and December 2011.
Sampling Method: Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
number of miscarriages | 2years
  The objective of this study was to evaluate the effect of three components: aspirin, alpha blockers and folic acid in women with miscarriages consecutive first-trimester mutation of the MTHFR C677T gene versus the effet of a combination of aspirin and folic acid in patients with three or more consecutive first-trimester miscarriages who were carrying the C677T MTHFR gene mutation

CONTACTS AND LOCATIONS:
Overall Officials: Moncef Ben Khlifa, MD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No